CLINICAL TRIAL: NCT02993185
Title: An Integrated Group-Individual Curriculum to Prevent Teen Pregnancy
Brief Title: Making Healthy Decisions: A Trial Evaluating the "Your Move" Teen Pregnancy-prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: ETR Associates (Other)
Responsible Party: Principal Investigator, Julie Downs, Associate Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000027
Record Dates: First submitted 2016-11-28; First posted 2016-12-15 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Pregnancy, Abdominal; Sexual Behavior; Sexually Transmitted Infection; Sexually Transmitted Diseases; Dietary Modification; Eating Behaviors
Keywords: pregnancy; adolescents; sexually transmitted diseases; decision making; prevention education
MeSH Terms: conditions — Pregnancy, Abdominal; Sexual Behavior; Sexually Transmitted Diseases; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Your Move (Experimental): Sex education intervention
  Interventions: Behavioral: Your Move
- Eat Smart (Active Comparator): Nutrition education intervention
  Interventions: Behavioral: Eat Smart

INTERVENTIONS:
Behavioral: Your Move — Your Move (YM) is an interactive sex education intervention. Groups of girls are randomly assigned to YM or Eat Smart (ES), a control interactive nutrition education intervention. Each program consist of seven 75-minute sessions, and each session contains 60 minutes of facilitator-led discussion, video clips, activities, and games as well as 15 minutes of "personal reflection" time during which girls practice the decision making skills they have learned. Participants complete online surveys about their attitudes, knowledge, and behavior related to food and nutrition and relationships and sex at baseline and also 3 months after the program ends.
  Arms: Your Move
Behavioral: Eat Smart — Eat Smart (ES) is an interactive nutrition education intervention. Groups of girls are randomly assigned to ES or Your Move, an interactive sex education intervention. Each program consist of seven 75-minute sessions, and each session contains 60 minutes of facilitator-led discussion, video clips, activities, and games as well as 15 minutes of "personal reflection" time during which girls practice the decision making skills they have learned. Participants complete online surveys about their attitudes, knowledge, and behavior related to food and nutrition and relationships and sex at baseline and also 3 months after the program ends.
  Arms: Eat Smart

SUMMARY:
The purpose of Making Healthy Decisions is to design and rigorously evaluate a new sexual health education program, "Your Move" (YM) against a nutrition control program, "Eat Smart" (ES). YM is intended to improve teen females' (ages 14-19) ability to make healthy sexual decisions with the ultimate goal of reducing unplanned pregnancies and STIs.

DETAILED DESCRIPTION:
Making Healthy Decisions includes two technology-based interventions designed to improve teen females' healthy decision making in relation to sexual relationships (YM) and nutrition (ES).

Health educators from Planned Parenthood are trained to implement both YM and ES at youth-serving community organizations in their geographic area across several U.S. states. In a multi-site randomized controlled trial, females ages 14-19 are recruited from their local community-based organization (CBO) into groups/cohorts of 8-12.

Each cohort is randomly assigned to participate in one of the two interventions prior to baseline data collection.

Participants attend seven 75-minute program sessions that include facilitator-led games, activities, and discussions as well as personal reflection time in which girls practiced healthy decision making individually on an electronic tablet.

Self-reported survey data related to attitudes, knowledge, and behavior around sex and nutrition are collected at baseline as well as 3 months after the intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* Female (or identify as female); age 14-19

Exclusion Criteria:

* Male (or identify as male); female older than 19 or younger than 14

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 808 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of sexual partners for vaginal intercourse | 3 months post intervention
  Number of partners with whom had vaginal sex
Number of incidents of vaginal sex without using hormonal contraception, copper IUD, or condoms | 3 months post intervention
  Number of times reported having vaginal sex without hormonal contraception, copper IUD, condoms, or insertive condoms
Number of incidents of vaginal sex without condoms | 3 months post intervention
  Number of times reported having vaginal sex without using condoms or insertive condoms

SECONDARY OUTCOMES:
Number of incidents of vaginal intercourse | 3 months post intervention
  Number of times had vaginal intercourse in the past 3 months
Condom errors or failure | 3 months post intervention
  Experienced any of 10 specific condom errors/failures during any condom use in the past 3 months (breakage, slippage, starting sex before putting condom on, removing condom before sex complete, open package with sharp object, use oil-based lubricant, put on condom before full erection, put on condom inside out and or flip it, had a problem that damaged condom & did not have another available, squeeze air from tip)
Number of incidents of vaginal, oral, or anal sex without using condoms | 3 months post intervention
  Number of times reported having vaginal, oral, or anal sex without using condoms or insertive condoms
Number of sexual partners for vaginal, oral, or anal intercourse | 3 months post intervention
  Number of partners with whom had vaginal, oral, or anal sex
Perceived self efficacy to communicate about sexual boundaries and condom use | 3 months post intervention
  Efficacy in communicating about sexual activity and condom use

OTHER OUTCOMES:
STI knowledge | 3 months post intervention
  Count of number of STI knowledge items correct out of 13.
Perceived self efficacy to use condoms | 3 months post intervention
  Perceived efficacy to get and use condoms.
Personal beliefs about what causes infertility | 3 months post intervention
  General beliefs about infertility/fear about ability to get pregnant.
Number of sexual partners without using condoms | 3 months post intervention
  Number of partners with whom had vaginal, oral, or anal sex without using condoms or insertive condoms
Birth control use | 3 months post intervention
  Use and consistency of use of 14 birth control methods (birth control pills, patch, Depo Provera, ring, IUD, implant, condoms, female condoms, diaphragm, cervical cap, sponge, spermicide, "safe time of month," "pull out"), and emergency contraception
Nutrition knowledge | 3 months post intervention
  Count of number of nutrition knowledge items correct out of 10.
Personal attitudes toward healthy eating | 3 months post intervention
  Mean score of 8 items on a 7 point scale on a newly developed questionnaire assessing healthy eating
Perceived self efficacy toward making healthy eating choices | 3 months post intervention
  Perceived efficacy to eat recommended number of servings of fruit and vegetables each day, avoid sugary drinks and eat breakfast daily
Nutrition behavior timeframe | 3 months post intervention
  Number of days report eating fruit, vegetables, too much food, not enough food, dining out, preparing meal at home, and eating breakfast
Nutrition behavior about quantity of fruit consumed | 3 months post intervention
  Amount (# of cups) of fruit consumed on a typical day
Nutrition behavior about quantity of vegetables consumed | 3 months post intervention
  Amount (# of cups) of vegetables consumed on a typical day
Nutrition behavior about quantity of sweetened beverage consumed | 3 months post intervention
  Amount (# of cups) of sweetened beverage consumed on a typical day
Nutrition behavior about food information when dining out | 3 months post intervention
  Notice or check nutrition information (on menu or online) when dining out
Nutrition behavior about food information when shopping | 3 months post intervention
  Notice or check nutrition information (food labels) when shopping

CONTACTS AND LOCATIONS:
Overall Officials: Julie Downs, PhD, Principal Investigator — Carnegie Mellon University; Pam Murray, MD, MHP, Principal Investigator — West Virginia University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Downs JS, Bruine de Bruin W, Fischhoff B, Murray PJ. Behavioral Decision Research Intervention Reduces Risky Sexual Behavior. Curr HIV Res. 2015;13(5):439-46. doi: 10.2174/1570162x13666150511145328. PMID 26149165
- [Result] Downs JS. Prescriptive scientific narratives for communicating usable science. Proc Natl Acad Sci U S A. 2014 Sep 16;111 Suppl 4(Suppl 4):13627-33. doi: 10.1073/pnas.1317502111. Epub 2014 Sep 15. PMID 25225369
- [Result] Downs JS, Murray PJ, Bruine de Bruin W, Penrose J, Palmgren C, Fischhoff B. Interactive video behavioral intervention to reduce adolescent females' STD risk: a randomized controlled trial. Soc Sci Med. 2004 Oct;59(8):1561-72. doi: 10.1016/j.socscimed.2004.01.032. PMID 15279915